CLINICAL TRIAL: NCT03010423
Title: An Interventional, Pilot Study to Evaluate the Efficacy of Oral Nicorandil on Improving Microvascular Function in Female Non-obstructive CAD Patients (SPET Study)
Brief Title: Efficacy Study of Oral Nicorandil on Improving Microvascular Function in Female Non-obstructive Coronary Artery Disease (CAD) Participants
Acronym: SPET
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated early, due to the lack of approval of data exportation from the Office of Human Genetic Resource Administration (OHGRA) China.
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono Co., Ltd., China (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR200505_506
Record Dates: First submitted 2017-01-03; First posted 2017-01-05 (Estimated); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Non-obstructive Coronary Artery Disease
Keywords: Non-obstructive coronary artery disease; Nicorandil
MeSH Terms: interventions — Nicorandil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nicorandil (Experimental)
  Interventions: Drug: Nicorandil

INTERVENTIONS:
Drug: Nicorandil — Participants received Nicorandil 5 milligram (mg) tablet, three times a day for 12 weeks.

SUMMARY:
The study is a single-center, interventional, pilot study to evaluate the improvement of microvascular function by positron emission tomography (PET) after twelve-week treatment of oral nicorandil in female non-obstructive CAD Participants.

ELIGIBILITY:
Inclusion criteria:

* Female
* Participants aged 18-70 years
* Participants with typical stable angina but without coronary obstruction (defined as coronary occlusion less than (<) 50%) by invasive coronary angiography or coronary computed tomography angiography (CTA) in recent three months
* All other long acting cardiovascular disease medicines, including but not limited to aspirin/clopidogrel, calcium channel blockers (CCB), Angiotensin-converting enzyme inhibitors (ACEI)/Angiotensin II Receptor Blockers (ARB), beta-blockers, statins, ivabradine, trimetazidine, et al, should be stable taken for at least two weeks before screening period
* For participants who met these four criteria above, MFR will be tested by stress PET. Participants whose MFR <3.0 could be included in the study

Exclusion criteria:

* Severe or uncontrolled hypertension (resting Systolic blood pressure [SBP] >=160 millimeter of mercury (mmHg), or resting Diastolic blood pressure [DBP] >=100mmHg at screening period)
* Participants with shock (including cardiogenic shock), or hypovolemia
* Severe hypotension (resting SBP<90mmHg，or resting DBP<60mmHg)
* Significant valvular heart disease, congenital heart disease or cardiomyopathy
* Congestive heart failure(New York Heart Association [NYHA] III-IV), echocardiographic ejection fraction<45%
* Acute pulmonary edema;
* Hepatic or renal dysfunction, defined as:

  * Serum Alanine Aminotransferase (ALT) > triple of the normal value upper limit;
  * Serum Aspartate Aminotransferase (AST) > triple of the normal value upper limit
  * Serum creatinine > twice of the normal value upper limit
* Glaucoma
* Active peptic ulcer or active skin ulcer
* Taking glyburide, phosphodiesterase type 5 (PDE-5) inhibitor, soluble guanylate cyclase stimulator(s)
* Known to be hypersensitivity to nicorandil, nitrates, niacin, or any of the excipient
* With contraindication to complete stress PET test
* No legal ability and legal ability is limited
* Participants unlikely to cooperate in the study or with inability or unwillingness to give informed consent
* Child-bearing period women without effective contraceptive measures, pregnancy and lactation
* Participation in another clinical trial within the past 30 days
* Other significant disease that in the Investigator's opinion would exclude the participant from the trial

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2019-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Serono Co., Ltd., China
Locations (1):
- Peking union medical college hospital, Beijing, China

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=EMR200505_506
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nicorandil
Started | 8
Completed | 0
Not Completed | 8
Not completed — Study termination | 8

BASELINE CHARACTERISTICS:
Arm/Group | Nicorandil
Number analyzed (Participants) | 8
Age, Customized [Number; unit: Participants] — The study was terminated early and due to the lack of approval of data exportation from the Office of Human Genetic Resource Administration (OHGRA) China, therefore the data could not be extracted and hence data reported here is as per the total range reflecting in the inclusion criteria.
  Participants
    Between >=18 and <= 70 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Myocardial Blood Flow Reserve (MFR) by Stress Positron Emission Tomography (PET) at Week 12
Description: Myocardial blood flow reserve is a measure of endothelial function measured by positron emission tomography.
Time Frame: Baseline, Week 12
Population: The study was terminated early and due to the lack of approval of data exportation from the Office of Human Genetic Resource Administration (OHGRA) China, the data could not be extracted. Therefore, no data available for the analyses.
Arm/Group | Nicorandil
Number analyzed (Participants) | 0

2. Secondary Outcome: Change From Baseline in Myocardial Blood Flow (MBF) by Rest Positron Emission Tomography (PET) at Week 12
Description: Myocardial blood flow is a measure of endothelial function measured by positron emission tomography.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Arm/Group | Nicorandil
Number analyzed (Participants) | 0

3. Secondary Outcome: Change From Baseline in Myocardial Blood Flow (MBF) by Stress Positron Emission Tomography (PET) at Week 12
Description: Myocardial blood flow is a measure of endothelial function measured by positron emission tomography.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Arm/Group | Nicorandil
Number analyzed (Participants) | 0

4. Secondary Outcome: Change From Baseline in Ejection Fraction at Week 12
Description: Echocardiography was used to measure ejection fraction.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Arm/Group | Nicorandil
Number analyzed (Participants) | 0

5. Secondary Outcome: Change From Baseline in Left Ventricular End-Systolic Dimension (LVESD) at Week 12
Description: Echocardiography was used to measure LVESD.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Arm/Group | Nicorandil
Number analyzed (Participants) | 0

6. Secondary Outcome: Change From Baseline in Left Ventricular Wall Thickness at Week 12
Description: Echocardiography was used to measure left ventricular wall thickness.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Arm/Group | Nicorandil
Number analyzed (Participants) | 0

7. Secondary Outcome: Change From Baseline in Cardiac Diastolic Function: Early [E] to Late [A] Ventricular Filling Velocities (E/A) Ratio at Week 12
Description: Echocardiography was used to measure E/A ratio.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Arm/Group | Nicorandil
Number analyzed (Participants) | 0

8. Secondary Outcome: Change From Baseline in Seattle Angina Questionnaire(SAQ) Score at Week 12
Description: Seattle angina questionnaire (SAQ) score will be classified into five dimensions: physical limitation (question 1), anginal stability (question 2), anginal frequency (question 3-4), treatment satisfaction (question 5-8) and disease perception (question 9-11). Individual dimensions of the SAQ are transformed into the standard score between 0 and 100. The range of scores was 0 to 100, with higher scores indicates better functioning.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Arm/Group | Nicorandil
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 15 months
Description: The study was terminated early and due to the lack of approval of data exportation from the Office of Human Genetic Resource Administration (OHGRA) China, the data could not be extracted. Thus, data for adverse event was not collected.
Arm/Group | Nicorandil
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The study was terminated early and due to the lack of approval of data exportation from the Office of Human Genetic Resource Administration (OHGRA) China, the data could not be extracted. Therefore, no data available for the analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-04-15): https://cdn.clinicaltrials.gov/large-docs/23/NCT03010423/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-13): https://cdn.clinicaltrials.gov/large-docs/23/NCT03010423/SAP_001.pdf